CLINICAL TRIAL: NCT06000774
Title: Ketogenic Diet in Eating Disorders to Target Metabolism and Normalize Persistent Eating Disorder Psychopathology
Brief Title: Therapeutic Ketogenic Diet in Anorexia Nervosa
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of California, San Diego (Other)
Responsible Party: Principal Investigator, Guido Frank, Professor, University of California, San Diego
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 807674
Record Dates: First submitted 2023-08-14; First posted 2023-08-21 (Actual); Last update posted 2025-09-05 (Actual); Status verified 2025-08

CONDITIONS: Anorexia Nervosa in Remission; Bulimia Nervosa; Anorexia Nervosa
MeSH Terms: conditions — Bulimia Nervosa; Anorexia Nervosa

STUDY DESIGN:
Intervention Model Description: Subjects will complete a 14-week therapeutic ketogenic diet (TKD)
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Therapeutic Ketogenic Diet (Experimental): A 2-week therapeutic ketogenic diet (TKD) induction will be implemented to establish nutritional ketosis (the goal are BHB blood levels of 0.5-3.0 millimoles per liter [mmol/L]). After establishing the ketotic state, study participants will continue TKD for 12 weeks.
  Interventions: Other: Therapeutic Ketogenic Diet

INTERVENTIONS:
Other: Therapeutic Ketogenic Diet — therapeutic ketogenic diet

SUMMARY:
This study will investigate the effects of therapeutic ketogenic diet (TKD) on eating behavior including drive to restrict, body dissatisfaction, mood and anxiety in individuals with anorexia nervosa who have been weight normalized (body mass index of 17.5 or greater) but continue to struggle with eating disorder behaviors including a high drive for thinness and body dissatisfaction.

The Underweight Anorexia Nervosa (AN) Sub-Study will investigate the effects of TKD on eating behavior including drive to restrict, body dissatisfaction, mood and anxiety in individuals with anorexia nervosa who are currently underweight (body mass index between 16.0 and 17.49) and continue to struggle with eating disorder behaviors including a high drive for thinness and body dissatisfaction.

The Bulimia Nervosa Pilot will will investigate the effects of TKD on eating behavior including drive to binge and purge, body dissatisfaction, mood and anxiety in individuals with bulimia nervosa.

DETAILED DESCRIPTION:
For this 14-week study, the investigator will recruit twenty individuals with anorexia nervosa who have been weight normalized but continue to have high impairment from the illness with a high (2 standard deviations above average) drive for thinness and body dissatisfaction and a high drive for food restriction and thus are at high risk for full relapse. Study participants will be carefully assessed and oriented to the ketogenic diet according to the procedures in our small previous trial (Calabrese, et al., 2022). The study will be conducted in a university medical environment, showing feasibility and safety in a typical medical setting. A commercial supplier will provide the ketogenic diet. After ketosis induction over two weeks, study participants will be assessed weekly for ketosis and mood, anxiety, and eating disorder symptoms.

For the BN Pillot study we will also complete a small pilot in 5 individuals with bulimia nervosa.

For the Underweight Anorexia Nervosa (AN) Sub-Study we will also recruit 30 individuals with anorexia nervosa who are mild to moderately underweight and have a body mass index of between 16.0 to 17.49.

Primary Objective 1 is to test the effects of ketogenic diet in individuals with anorexia nervosa who are weight recovered but continue to suffer severely from drive for thinness and are at very high relapse risk. Participants will be evaluated for tolerability of the study and weight trajectory. Primary Objective 2 is to assess improvement in AN symptoms and behaviors in relation to the ketogenic diet over a 12-week course. Participants will be assessed for specific symptoms such as drive for thinness and body dissatisfaction, fear of eating and weight gain. Primary Objective 3 is to assess the underlying genetic basis for the treatment effect of the ketogenic diet.

Bulimia Nervosa Pilot Objective 1: To test the effects of ketogenic diet in individuals with bulimia nervosa.

Bulimia Nervosa Pilot Objective 2: To assess improvement in BN symptoms and behaviors in relation to the ketogenic diet over a 2-week induction period followed by a 12-week course of the intervention. We expect especially a reduction in binge eating episodes and associated purging episodes in response to the treatment and in addition to improvement of the cognitive emotional symptoms.

Underweight AN Sub-Study Objective 1: To test the effects of ketogenic diet in individuals with anorexia nervosa who are currently mildly underweight and assess how the intervention impacts weight normalization in this population.

Underweight AN Sub-Study Objective 2: To assess improvement in AN symptoms and behaviors in relation to the ketogenic diet over a 2-week induction period followed by a 12-week course of the intervention.

Underweight AN Sub-Study Objective 3: To assess the underlying genetic basis for the treatment effect of the ketogenic diet.

ELIGIBILITY:
Weight-Recovered AN Inclusion Criteria:

1. Provision of signed and dated informed consent form
2. Stated willingness to comply with all study procedures and availability for the duration of the study
3. Persons, aged 18 to 45 years
4. History of anorexia nervosa according to DSM-5 criteria
5. Weight recovered at the time of study inclusion (body mass index > 17.5 kg/m2)
6. Greater or equal to 2 standard deviations scores of eating disorder-relevant behaviors on the Eating Disorder Inventory-3 and Eating Disorder Examination Questionnaire
7. The following types of psychiatric medications are allowed: antidepressant, anxiolytic, atypical antipsychotic, mood stabilizers
8. English is primary spoken language

Weight-Recovered AN Exclusion Criteria:

1. Pregnancy or lactation
2. Electrolyte, blood count, kidney function or liver function abnormalities
3. Psychosis
4. Neurocognitive disorders including dementias or traumatic brain injury that is symptomatic
5. Current alcohol use disorder (AUD) or substance use disorder (SUD) according to DSM-5 criteria
6. Uncontrolled hypertension
7. Hepatic impairment (Class-Pugh b or c)
8. Diabetes mellitus
9. Family history of porphyria
10. History of recent heart attack, vascular disease, or any other current acute medical conditions as determined by the principal investigator
11. Inability or unwillingness to adhere to the TKD diet for the duration of the study
12. Blind or illiterate individuals

Underweight AN Sub-Study Inclusion Criteria:

1. Provision of signed and dated informed consent form
2. Stated willingness to comply with all study procedures and availability for the duration of the study
3. Persons, aged 18 to 45 years
4. Anorexia nervosa according to DSM-5 criteria
5. Current Body Mass Index (BMI) at the time of study inclusion of 16.0 to 17.49
6. An elevated EDE-Q global score of 2.09 or greater
7. The following types of psychiatric medications are allowed: antidepressant, anxiolytic, atypical antipsychotic, mood stabilizers
8. English is primary spoken language

Underweight AN Sub-Study Exclusion Criteria:

1. Pregnancy or lactation
2. Electrolyte, blood count, kidney function or liver function abnormalities
3. Psychosis
4. Neurocognitive disorders including dementias or traumatic brain injury that is symptomatic
5. Current alcohol use disorder (AUD) or substance use disorder (SUD) according to DSM-5 criteria
6. Uncontrolled hypertension
7. Hepatic impairment (Class-Pugh b or c)
8. Diabetes mellitus
9. Family history of porphyria
10. History of recent heart attack, vascular disease, or any other current acute medical conditions as determined by the principal investigator
11. Inability or unwillingness to adhere to the TKD diet for the duration of the study
12. Blind or illiterate individuals

Bulimia Nervosa Pilot Inclusion Criteria:

1. Provision of signed and dated informed consent form
2. Stated willingness to comply with all study procedures and availability for the duration of the study
3. Persons, aged 18 to 45 years
4. History of bulimia nervosa according to DSM-5 criteria
5. An elevated EDE-Q global score of 2.09 or greater
6. The following types of psychiatric medications are allowed: antidepressant, anxiolytic, atypical antipsychotic, mood stabilizers
7. English is primary spoken language

Bulimia Nervosa Pilot Exclusion Criteria:

1. Pregnancy or lactation
2. Electrolyte, blood count, kidney function or liver function abnormalities
3. Psychosis
4. Neurocognitive disorders including dementias or traumatic brain injury that is symptomatic
5. Current alcohol use disorder (AUD) or substance use disorder (SUD) according to DSM-5 criteria
6. Uncontrolled hypertension
7. Hepatic impairment (Class-Pugh b or c)
8. Diabetes mellitus
9. Family history of porphyria
10. History of recent heart attack, vascular disease, or any other current acute medical conditions as determined by the principal investigator
11. Inability or unwillingness to adhere to the TKD diet for the duration of the study
12. Blind or illiterate individuals

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 20 (Estimated)
Dates: Start 2023-10-03 (Actual); Primary Completion 2027-06 (Estimated); Study Completion 2027-06-30 (Estimated)

PRIMARY OUTCOMES:
To assess the safety and tolerability in individuals with anorexia nervosa who are weight recovered, individuals with anorexia nervosa who are currently underweight, and individuals with bulimia nervosa using weekly body weight measurements. | Weekly for the duration of the study intervention (14 weeks)
  Weekly weights will be obtained to assess whether subjects remain within a normal weight range.
To assess the safety and tolerability in individuals with anorexia nervosa (AN) who are weight recovered, AN individuals who are currently underweight, and Bulimia Nervosa individuals using the Committee of Clinical Investigations UKU-Side Effect Scale | At weeks 4, 8, 12, 14
  The UKU assesses psychiatric, neurologic, autonomic, and other side effects.
Measurement of drive for weight loss, fear of weight gain and body image distortion using the Eating Disorder Examination Questionnaire (EDEQ) Global Score, EDEQ Eating Restraint Score, and EDEQ Weight Concern | At baseline, Week 1, 2, 3, 4, 5, 6, 7, 8, 9, 10, 11, 12, 13, 14, 3 month follow-up
  The Eating Disorders Examination Questionnaire a self report assessment that measures core eating disorder symptoms. Subjects will complete this measure at the beginning and end of the study and weekly throughout the 14-week intervention and the investigator will measure the change in scores. The EDE Global, Eating Restraint, and Weight Concern scales have a range of 0 to 6 where higher scores mean worse outcome.
Measurement of the relationship between genotype and improvement of eating disorder symptoms | At baseline
  In order to identify potential genetic signatures that may predict response to treatment, Whole Exome Sequencing will be conducted on participants.

CONTACTS AND LOCATIONS:
Overall Officials: Guido Frank, MD, Principal Investigator — University of California, San Diego
Locations (1):
- University of California San Diego, San Diego, California, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Scolnick B, Zupec-Kania B, Calabrese L, Aoki C, Hildebrandt T. Remission from Chronic Anorexia Nervosa With Ketogenic Diet and Ketamine: Case Report. Front Psychiatry. 2020 Jul 30;11:763. doi: 10.3389/fpsyt.2020.00763. eCollection 2020. PMID 32848935
- [Background] Frank GKW, Shott ME, DeGuzman MC. The Neurobiology of Eating Disorders. Child Adolesc Psychiatr Clin N Am. 2019 Oct;28(4):629-640. doi: 10.1016/j.chc.2019.05.007. Epub 2019 Jul 4. PMID 31443880
- [Background] Frank GKW, Shott ME, Stoddard J, Swindle S, Pryor TL. Association of Brain Reward Response With Body Mass Index and Ventral Striatal-Hypothalamic Circuitry Among Young Women With Eating Disorders. JAMA Psychiatry. 2021 Oct 1;78(10):1123-1133. doi: 10.1001/jamapsychiatry.2021.1580. PMID 34190963
- [Background] Dignon A, Beardsmore A, Spain S, Kuan A. 'Why I won't eat': patient testimony from 15 anorexics concerning the causes of their disorder. J Health Psychol. 2006 Nov;11(6):942-56. doi: 10.1177/1359105306069097. PMID 17035265
- [Background] Calabrese L, Scolnick B, Zupec-Kania B, Beckwith C, Costello K, Frank GKW. Ketogenic diet and ketamine infusion treatment to target chronic persistent eating disorder psychopathology in anorexia nervosa: a pilot study. Eat Weight Disord. 2022 Dec;27(8):3751-3757. doi: 10.1007/s40519-022-01455-x. Epub 2022 Aug 23. PMID 35997954